CLINICAL TRIAL: NCT00202618
Title: The Reduction of Microalbuminuria in Japanese Hypertensive Subjects With Type 2 Diabetes Mellitus Treated With Valsartan or Amlodipine: Study Design for the Shiga Microalbuminuria Reduction Trial (SMART)
Brief Title: Rationale and Design for Shiga Microalbuminuria Reduction Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiga University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2005-07

CONDITIONS: Hypertension; Diabetes Mellitus; Albuminuria
Keywords: Hypertension; Type 2 diabetes mellitus; Microalbuminuria; Amlodipine; Calcium channel blocker; Valsartan; Angiotensin type 2 receptor blocker
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Albuminuria; Diabetes Mellitus, Type 2 | interventions — Valsartan; Amlodipine

INTERVENTIONS:
Drug: Valsartan
Drug: Amlodipine

SUMMARY:
The purpose of this trial are to evaluate the reduction of urinary albumin excretion by an angiotensin receptor blocker (ARB), valsartan, in comparison with a calcium channel blocker (CCB), amlodipine, in Japanese hypertensive patients with type 2 diabetes mellitus and microalbuminuria under strict blood pressure control, and to compare the additional effects of an ARB or a CCB in combination with angiotensin-converting enzyme (ACE) inhibitor treatment.

DETAILED DESCRIPTION:
Microalbuminuria in diabetic patients is an established risk marker for the progression of diabetic nephropathy and for cardiovascular mortality. Intervention trials have demonstrated that drugs that blockade the renin-angiotensin system can reduce microalbuminuria in Caucasian patients with type 2 diabetes mellitus and microalbuminuria, regardless of blood pressure level. However, it remains uncertain whether angiotensin receptor blockers or calcium channel blockers give a greater reduction of microalbuminuria. The Shiga Microalbuminuria Reduction Trial (SMART) is a prospective, multicentre, randomized, active-controlled, two-arm parallel treatment group comparison study aimed at evaluating reduction of microalbuminuria in 160 Japanese hypertensive patients with type 2 diabetes mellitus and microalbuminuria. The trial consists of an 8-week observation period for screening and washout, and a 24-week intervention period. After the observation period, patients are randomized to either amlodipine 5 mg once daily or valsartan 80 mg once daily as an initial dose. After four weeks, if patients cannot achieve the target blood pressure (<130/80 mmHg) with the initial dose of a study drug, doses are titrated up to amlodipine 10 mg once daily or valsartan 160 mg once daily. The primary endpoints are a change in the rate of urinary albumin excretion from baseline, a normalization of microalbuminuria, and a 50% reduction in urinary albumin excretion from baseline, which are compared between treatment groups. This study will provide additional data for the treatment of hypertension and microalbuminuria and has important health care implications for Japanese patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patient with type 2 diabetes
* Microalbuminuria defined as a urinary albumin excretion of 30 to 300 mg/gCr

Exclusion Criteria:

* Type 1 diabetes mellitus
* Pregnant women and women of childbearing potential
* Severe hypertension (> 180/110 mmHg), malignant hypertension, secondary hypertension
* History of cardiovascular diseases in the preceding 6 months (including symptomatic heart failure, unstable angina, myocardial infarction, the performance of percutaneous transluminal coronary angioplasty [PTCA], or coronary artery bypass graft [CABG], severe arrhythmia, or second or third degree atrioventricular [AV] block)
* History of clinically significant valvular disease (e.g., aortic stenosis, mitral insufficiency)
* History of cerebral infarction, cerebral hemorrhage, or transient ischemic attack
* Serum creatinine level >1.5 mg/dl
* Persistent hematuria
* Serum potassium > 5.6 mEq/L (hyperkalemia)
* Severe hepatic disorder (e.g., hepatic failure, hepatic cirrhosis)
* Complication of an allergy of potential clinical concern
* Hypersensitivity to ARBs or CCBs
* Gastrointestinal surgery or gastrointestinal disorders which could interfere with drug absorption
* Autoimmune disease
* Participation in any intervention trial within 3 months prior to the observation period
* Patients who are unwilling or unable to comply with the trial protocol
* Concomitant use of other ARBs, CCBs, or potassium-retaining diuretics

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2003-12; Study Completion 2006-06

PRIMARY OUTCOMES:
A change in the rate of urinary albumin excretion (UAE) from the baseline to the end of study
A normalization of microalbuminuria (normoalbuminuria)
A 50% reduction in UAE from the baseline

SECONDARY OUTCOMES:
A change in urinary type IV collagen from the baseline to the end of the intervention period
A change in high sensitivity C-reactive protein (hsCRP) from the baseline to the end of the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Atsunori Kashiwagi, Professor, Study Chair — Shiga University of Medical Science
Locations (1):
- Shiga University of Medical Science, Ōtsu, Shiga, Japan

REFERENCES:
- [Derived] Shiga Microalbuminuria Reduction Trial (SMART) Group; Uzu T, Sawaguchi M, Maegawa H, Kashiwagi A. Impact of renin-angiotensin system inhibition on microalbuminuria in type 2 diabetes: a post hoc analysis of the Shiga Microalbuminuria Reduction Trial (SMART). Hypertens Res. 2008 Jun;31(6):1171-6. doi: 10.1291/hypres.31.1171. PMID 18716365 (Retraction: PMID 24671017 Hypertens Res. 2014 Jun;37(6):598)